CLINICAL TRIAL: NCT07399002
Title: Long Coronary Lesions: Safety and Performance of the Ultimaster Nagomi™ Stent in This Setting With a One-to-one Approach -One Lesion, One Stent- LONG NAGOMI™ PMCF STUDY
Brief Title: LONG NAGOMI™ PMCF STUDY
Acronym: LONG NAGOMI
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: rEPIC19- LONG NAGOMI
Record Dates: First submitted 2025-11-24; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up)
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: LONG NAGOMI

INTERVENTIONS:
Device: LONG NAGOMI — Patients in whom treatment with long nagomi has been attempted

SUMMARY:
The study is designed as a prospective, multi-center, observational PMCF (post-market clinical follow-up) study of the Ultimaster Nagomi™ _stent (lengths of 38, 44 and 50 mm) in the treatment of coronary artery disease according to the indications approved in the CE marking.

DETAILED DESCRIPTION:
The study serves to fulfill post marketing surveillance requirements for the Ultimaster Nagomi™ stent. This is a PMCF study of real-world use of the Ultimaster Nagomi™ DES aimed to reaffirm the device claims of effectiveness and safety, no comparator is required to meet these specified objectives and endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet ALL inclusion criteria will be included:
* Patients aged ≥ 18 years AND;
* Patients who according to standard practice of the hospital are amenable to PCI as indicated and considered adequate according to the European clinical practice guidelines on coronary revascularization AND;
* Patients with at least one lesion fulfilling the "long lesion criteria" suitable for a single stent approach AND;
* Patients who have been informed of the characteristics of the study and have provided written informed consent AND;
* Intention to treat all lesions with the Ultimaster Nagomi™ stent

Exclusion Criteria:

* Patients must not meet any of the following exclusion criteria:
* Patients who expressly decline to participate in the study.
* Pregnant or breastfeeding women.
* Patients with acute coronary syndrome (ACS) under conditions of cardiogenic shock (Killip class 4).
* Patients with contraindications or hypersensitivity to sirolimus.
* Patients with a life expectancy of less than 2 years.
* Patients in whom any surgery requiring general anesthesia is planned, comorbidity or indication likely necessitating the discontinuation of dual anti-platelet therapy before the recommended duration of dual anti-platelet therapy per the ESC or national guidelines.
* Patients included in other clinical trials that did not reach the primary objective.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PCI with implantation of a Long Nagomi stent
Sampling Method: Non-Probability Sample
Enrollment: 1039 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 1 year
  Target Lesion Failure defined as the composite of cardiovascular death, target-vessel related myocardial infarction and clinically driven target lesion revascularization at 1-year post-procedure.

SECONDARY OUTCOMES:
Device success | Periprocedural
  Device success defined as delivery success (achievement of successful delivery of study stent to the target lesion, expansion of the study stent and withdrawal of the delivery catheter) with a final residual diameter stenosis of the target lesion of < 20% by visual assessment and/or < 30% by QCA, using the assigned device only.
Safety of the stent: Freedom from Accidental dislodgement of the stent | Periprocedural
  Safety of the stent defined as an absence of Accidental stent dislodgement
Safety of the stent: Freedom from Balloon rupture | Periprocedural
  Safety of the stent defined as an absence of Balloon rupture o Hypotube rupture.
Safety of the stent: Freedom from Hypotube rupture o Hypotube rupture | Periprocedural
  Safety of the stent defined as an absence of o Hypotube rupture o Hypotube rupture.
Safety of the procedure: Freedom from Challenging withdrawal | Periprocedural
  Safety of the procedure defined as an absence of Challenging withdrawal
Safety of the procedure: Freedom from coronary perforation | Periprocedural
  Safety of the procedure defined as an absence of coronary perforation
Safety of the procedure: Freedom from dissection >C | Periprocedural
  Safety of the procedure defined as an absence of dissection >C
Safety of the procedure: Freedom from no-reflow | Periprocedural
  Safety of the procedure defined as an absence of no-reflow
Safety of the procedure: Freedom from stent thrombosis | Periprocedural
  Safety of the procedure defined as an absence stent thrombosis
Procedure success | Periprocedural
  To assess the procedure success rate defined as the achievement of < 20% residual stenosis by visual assessment in all target lesions using any percutaneous method without the occurrence of death, Q wave or WHO defined non-Q wave myocardial Infarction, or need for new revascularization of the target lesion during the hospital stay.
Performance of the Ultimaster Nagomi™ stent in Severe calcified lesions | Periprocedural
  To assess Performance of the Ultimaster Nagomi™ stent in Severe calcified lesions
Performance of the Ultimaster Nagomi™ stent in Severe tortuous vessels | Periprocedural
  To assess Performance of the Ultimaster Nagomi™ stent in Severe tortuous vessels
Performance of the Ultimaster Nagomi™ stent in Distal vessels | Periprocedural
  To assess Performance of the Ultimaster Nagomi™ stent in Distal vessels
Angina status assessment Seattle Angina Questionnaire (SAQ) | Baseline
  Angina status assessment Seattle Angina Questionnaire (SAQ)
Angina status assessment Seattle Angina Questionnaire (SAQ) | 12 monts
  Angina status assessment Seattle Angina Questionnaire (SAQ)
Quality of Life assessed as per EuroQl five-dimensional (EQ-5D) questionnaire | After PCI
  Quality of Life assessed as per EuroQl five-dimensional (EQ-5D) questionnaire
Quality of Life assessed as per EuroQl five-dimensional (EQ-5D) questionnaire | 12 Months
  Quality of Life assessed as per EuroQl five-dimensional (EQ-5D) questionnaire
Cardiovascular death | 12 months
  Percentage of cardiovascular death
Target-vessel related myocardial infarction | 12 Months
  Percentage of target-vessel related myocardial infarction
Clinically driven target lesion revascularization | 12 months
  Percentage of clinically driven target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario Marqués de Valdecilla, Santander

REFERENCES:
- [Background] Khan, M. (2024). Prevalence of in-stent restenosis in patients having drug eluting stents with lengths exceeding 40mm: a single-center study. JHRR, 4(2), 837-841. doi.org/10.61919/jhrr.v4i2.960
- [Background] Khanal S, Agarwal A, Kumar B. One-Year Outcomes of Long Coronary Drug-Eluting Stents (>/=40 MM) in Patients With Diffuse Coronary Artery Disease: Findings From a Tertiary Care Hospital in North India. Cureus. 2024 May 3;16(5):e59611. doi: 10.7759/cureus.59611. eCollection 2024 May. PMID 38832189
- [Background] Park KE, Wu CJ, Chehab B, Maksoud A, Bertolet B, Ying SW, Simoes T, Pingle SC, Chang CJ. One-year Outcomes of XIENCE Skypoint 48-mm Drug-Eluting Stents in Long Coronary Lesions: The SPIRIT 48 Trial. J Soc Cardiovasc Angiogr Interv. 2023 May 18;2(4):101001. doi: 10.1016/j.jscai.2023.101001. eCollection 2023 Jul-Aug. PMID 39131646
- [Background] Patra S, Chakraborty RN, Pande A, Banerjee S, Jena M, Mandal PC, De SK, Khan A, Das SS, Ghosh D, Nag R. Zotarolimus-eluting Resolute Integrity versus everolimus-eluting Xience Xpedition stents in the management of very long (>30mm) de novo coronary artery stenosis. Cardiovasc Revasc Med. 2017 Apr-May;18(3):160-164. doi: 10.1016/j.carrev.2016.12.007. Epub 2016 Dec 15. PMID 28017259
- [Background] Gautier A, Hovasse T, Arroyo D, Unterseeh T, Garot P, Champagne S, Neylon A, Sanguineti F, Benamer H, Chevalier B, Lefevre T. Safety and efficacy of 48 mm Xience Xpedition everolimus-eluting stent for the treatment of long coronary lesions. Catheter Cardiovasc Interv. 2022 Aug;100(2):179-187. doi: 10.1002/ccd.30249. Epub 2022 May 27. PMID 35621281